CLINICAL TRIAL: NCT05594121
Title: A Pragmatic, Multi-centre, Open-label, Randomized, 12-month, Parallel Group, Superiority Study to Compare the Effectiveness of Subcutaneous Buprenorphine Depot (Sublocade®) vs Daily Sublingual Buprenorphine With Naloxone (Suboxone®) for the Treatment of Opioid Use Disorder
Brief Title: Monthly Versus Daily Buprenorphine Formulations for Treatment of Opiate Use Disorder
Acronym: STOPIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Giulio DiDiodato, Chief Research Scientist, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R22-004
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Moderate to Severe Opioid Use Disorder
MeSH Terms: interventions — Sublocade; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: Pragmatic, multi-centre, randomised, controlled, open-label, superiority study with two parallel groups and primary endpoints of opioid positivity and healthcare utilization at 12 months after enrollment. Randomization will be performed with a 1:1 allocation ratio using a stratified, permuted-block group schema according to the following strata (no fixed ratio):
  1. RAAM clinic site (Barrie, Orillia, Midland, Wasaga Beach)
  2. Severity of OUD according to DSM-V criteria (moderate vs severe)
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded to intervention code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended-release subcutaneous buprenorphine (SC-BPN-XR) (Experimental): For eligible patients randomly allocated to SC-BPN-XR, the first dose will be administered at the time of randomization (Day 0). SC-BPN-XR comes in two formulations, 100 mg and 300 mg buprenorphine doses in a pre-filled syringe. SC-BPN-XR administration is by subcutaneous injection in the abdomen. SC-BPN-XR is administered at intervals ≥26 days. For patients randomly allocated to SC-BPN-XR, they will receive the 300 mg dose for the first 2 months, followed by the 100 mg dose every month until the end of the 12-month period. All SC-BPN-XR doses will be administered in clinics by trained personnel. All patients receiving SC-BPN-XR will have their vital signs monitored every 5 minutes for 15 minutes after the injection before leaving the clinic.
  Interventions: Drug: Extended Release Subcutaneous Buprenorphine
- Immediate-release sublingual buprenorphine/naloxone (SL-BPN/NX) (Active Comparator): For eligible patients randomly allocated to SL-BPN/NX, the first study dose will be administered at the time of randomization (Day 0) and will match the SL-BPN/NX type (tablet versus film), route (sublingual versus buccal) and dose used for stabilization prior to study enrollment. For the first 2 weeks of the study period, all SL-BPN/NX administration will be directly observed at community pharmacies by trained personnel according to the usual standard of care. Subsequent to this period, healthcare providers and participants will develop a care plan for ongoing directly observed therapy vs unsupervised take-home dosing according to usual standard of care.
  Interventions: Drug: Immediate Release Sublingual Buprenorphine

INTERVENTIONS:
Drug: Extended Release Subcutaneous Buprenorphine — Monthly subcutaneous injections of long-acting buprenorphine
  Other Names: Sublocade
  Arms: Extended-release subcutaneous buprenorphine (SC-BPN-XR)
Drug: Immediate Release Sublingual Buprenorphine — Daily sublingual fast-acting buprenorphine
  Other Names: Suboxone
  Arms: Immediate-release sublingual buprenorphine/naloxone (SL-BPN/NX)

SUMMARY:
Opioid use disorder and opioid-related deaths are increasing across Canada. The mainstay of medical treatment includes either full (methadone) or partial (buprenorphine) opioid agonist therapy. In Canada, there are 2 buprenorphine formulations, an immediate-release (Suboxone) and extended-release(Sublocade). These treatments have been shown to be equivalent for medication adherence and treatment retention. However, Sublocade costs 8-times more, and 50% of patients must pay out-of-pocket if they prefer this treatment option. This study is needed to demonstrate the superior benefits of Sublocade on important clinical outcomes to demonstrate its cost-effectiveness and justify expanded insured access across Canada.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) as a "problematic pattern of opioid use leading to clinically significant impairment or distress." The DSM-V also uses the number of criteria present to categorize the severity of OUD, with mild OUD defined as having 2-3 criteria present, moderate OUD defined as having 4-5 criteria present, and severe OUD defined as having ≥6 criteria present. Opioid use disorder and opioid-related deaths are increasing in Ontario and Canada. Compared to 2016, the age-adjusted opioid-related mortality rates in 2020 have increased by 161% in Ontario to 16.5 per 100 000 population and 114% in Canada to 16.7 per 100 000 population. Like deaths, opioid-related healthcare utilization as measured by hospitalization and emergency department visits have also been increasing over the same time period. Compared to 2016, the age-adjusted opioid-related hospitalization rates in 2020 have increased by 19.8% in Ontario to 16.3 per 100 000 population and 5.9% in Canada to 17.8 per 100 000 population. Emergency room visits have increased by 166% during the same time period in Ontario to 84.5 per 100 000 population. The median length of hospitalization from 2016 to 2020 has remained unchanged at 3 days (Range 1 to 207 days), with an average cost per hospitalization of $9 626 (CDN) (Range $26 to $296 831). Opiate substitution treatment with either full (methadone) or partial (buprenorphine) opioid agonist therapy (OAT) has been shown to reduce self-reported opioid use or opiate positive urine drug tests compared to detoxification or psychological treatments. There are 2 main opioid agonists used to treat OUD, methadone and buprenorphine. Buprenorphine has been approved by Health Canada for use in OUD, and is available in immediate (Suboxone®) and extended-release (Sublocade®) formulations. Monthly subcutaneous buprenorphine (SC-BPN-XR) has been shown to be non-inferior to daily sublingual buprenorphine/naloxone (SL-BPN/NX) for medication adherence and treatment retention. The Canadian pharmaceutical costs of Sublocade® and Suboxone® differ substantially , with monthly costs for Sublocade 8-fold higher than Suboxone. The majority of patients meeting criteria for Sublocade® use must pay for the drug out-of-pocket resulting in significant restriction to access for this population that has a high burden of chronic homelessness and poverty. A recent pharmacoeconomic report by the Canadian Agency for Drugs and Technologies in Health (CADTH) concluded that the current evidence base for supporting cost-effectiveness of Sublocade® over Suboxone is limited by the absence of studies directly comparing the effectiveness of the two treatments on clinically important outcomes such as healthcare utilization. With limited evidence and significant uncertainty, the CADTH analysis suggested that a price reduction of at least 73% would be required for Sublocade® to be a cost-effective alternative to Suboxone. A real-world (pragmatic) randomised study is therefore needed to compare the treatment effectiveness of Sublocade® versus Suboxone® in Canadian patients attending RAAM clinics for OAT for moderate- to severe-OUD. This study is needed to demonstrate the superior benefits of Sublocade® on important clinical outcomes such as reduced opioid and healthcare utilization in order to demonstrate its cost-effectiveness and justify expanded access for this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65 years old
* OAT indicated for moderate- to severe-OUD
* Attend a RAAM clinic in the North Simcoe Muskoka Local Health Integrated Network for opiate substitution treatment
* Successfully completed induction and stabilization OAT with Suboxone® tablet or film defined as receiving 8mg/2mg to 24mg/6mg of Suboxone® for ≥7 days with no evidence of allergic reaction to Suboxone®, Clinical Opiate Withdrawal Scale (COWS) score ≤12 (scale:0-48) for ≥24 hours, and Opiate Craving Visual Analog Scale (VAS) score ≤20 (scale:0-100)) for ≥24 hours
* Must have an active Ontario Health Insurance Plan number
* Must have a telephone that can receive calls, text messages or emails
* Must have drug insurance coverage for either medication for duration of study or demonstrate ability to pay for the drug out-of-pocket

Exclusion Criteria:

* Receiving any investigational drug for OUD in previous 4 weeks
* Congenital long QTc syndrome or QTc prolongation at baseline by electrocardiogram (QTc ≥450 milliseconds in men and QTc ≥470 milliseconds in women)
* Pregnant or lactating women
* Women of childbearing potential who are not using an effective and reliable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Opioid positivity | every 7 days for 12 months
  Difference in proportions of relapse-free weeks (RFWs) at 12-months from the date of randomization, where relapse-free weeks are defined by the cumulative number of weeks alive during the study period in which there was a negative urine drug screen and negative self-report for non-prescribed opioids. The potential number of RFWs for each patient is the cumulative number of weeks that the patient is alive during the 12-month study period, with a maximum of 48 weeks. A week is defined as a consecutive 7-day period starting on the day of the week that randomization occurred.
Healthcare utilization | 12 months
  Difference in incidence rates of healthcare days at 12-months from the date of randomization, where healthcare days represent the number of days alive and registered for an emergency room visit or admitted to an acute care or mental health facility for opioid-related harms or poisonings. For each group, the incidence rate is calculated by dividing the total number of healthcare days by the total person days exposure over the study period. The potential number of healthcare days for each patient is the number of days alive during the 12-month study period, with the maximum being 365 days. Any day in which a patient is documented to have had an emergency room visit or is admitted to an acute care or mental health facility for any opioid-related harm or poisoning will be counted as a healthcare day. Only those healthcare days in which opioid use was considered to be influential to the ER visit or hospitalization will be included in the final analysis.

SECONDARY OUTCOMES:
Medication Satisfaction | Every 6 weeks starting on week 6 after randomization for 12 months
  Difference in the Medication Satisfaction Questionnaire scores. The questionnaire is a single-item, global, patient-completed instrument that has been validated to measure treatment satisfaction, initially in patients receiving antipsychotic treatment for schizophrenia, but subsequently used in trials measuring satisfaction with opiate substitution treatment. The question will be read aloud by the RAAM clinic healthcare providers or study personnel to the patient. The question asks, "Overall, how satisfied are you with your current Suboxone®/Sublocade® medication?". The responses are on a 7-point Likert scale, ranging from 1=extremely dissatisfied to 7=extremely satisfied.
Quality of Life Score | At time of randomization (baseline), then week 12, week 24 and week 36
  Difference in the World Health Organization Quality of Life - BREF scores (WHOQOL-BREF). The 26-item questionnaire is a validated, self-report instrument that assesses 4 domains of quality of life: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). There are also 2 items that measure overall quality of life and general health. The questionnaire takes 15-20 minutes to complete. The questionnaire prefaces each item, "Think about your life in the last two weeks..". The responses are on a 5-point Likert scale, ranging from 1=not at all/very dissatisfied/never/very poor to 5=very good/very satisfied/an extreme amount/extremely/completely/always, depending on the item.
Clinic Retention | 12 months
  Difference in proportion of patients who attend ≥80% of scheduled clinic visits, where a clinic visit is defined as a scheduled visit with a RAAM clinic healthcare provider for any reason, including urine drug testing, medication administration, or counselling. The number of clinic visits any patient will be assigned will include those scheduled as part of the trial and any other visits scheduled at the discretion of the RAAM clinic healthcare providers.
Mortality | 12 months
  Difference in mortality proportions, where mortality is defined as any death attributable to opioid use regardless of the intent.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wong, MN, Principal Investigator — Royal Victoria Regional Health Centre; Giulio DiDiodato, PhD, Principal Investigator — Royal Victoria Regional Health Centre
Locations (5):
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - RAAM Clinic (Barrie), Barrie, Ontario
  - RAAM Clinic (Midland0, Midland, Ontario
  - RAAM Clinic (Orillia), Orillia, Ontario
  - RAAM Clinic (Wasaga Beach), Wasaga Beach, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders (5th ed.). (American Psychiatric Publishing, Inc., 2013).
- [Background] Ontario Agency for Health Protection and Promotion. Opioid mortality surveillance report: analysis of opioid-related deaths in Ontario July 2017-June 2018. (2019).
- [Background] Special Advisory Committee on the Epidemic of Opioid Overdoses. Opioid and Stimulant-related Harms in Canada. https://health-infobase.canada.ca/substance-related-harms/opioids-stimulants/ (2021).
- [Background] Public Health Ontario. Opioid-related Morbidity and Mortality in Ontario. https://www.publichealthontario.ca/en/data-and-analysis/substance-use/interactive-opioid-tool#/trends (2021).
- [Background] Nielsen S, Larance B, Degenhardt L, Gowing L, Kehler C, Lintzeris N. Opioid agonist treatment for pharmaceutical opioid dependent people. Cochrane Database Syst Rev. 2016 May 9;(5):CD011117. doi: 10.1002/14651858.CD011117.pub2. PMID 27157143
- [Background] Bruneau J, Ahamad K, Goyer ME, Poulin G, Selby P, Fischer B, Wild TC, Wood E; CIHR Canadian Research Initiative in Substance Misuse. Management of opioid use disorders: a national clinical practice guideline. CMAJ. 2018 Mar 5;190(9):E247-E257. doi: 10.1503/cmaj.170958. No abstract available. PMID 29507156
- [Background] Sordo L, Barrio G, Bravo MJ, Indave BI, Degenhardt L, Wiessing L, Ferri M, Pastor-Barriuso R. Mortality risk during and after opioid substitution treatment: systematic review and meta-analysis of cohort studies. BMJ. 2017 Apr 26;357:j1550. doi: 10.1136/bmj.j1550. PMID 28446428
- [Background] Bahji A, Cheng B, Gray S, Stuart H. Reduction in mortality risk with opioid agonist therapy: a systematic review and meta-analysis. Acta Psychiatr Scand. 2019 Oct;140(4):313-339. doi: 10.1111/acps.13088. PMID 31419306
- [Background] Galanter M, Femino J, Hunter B, Hauser M. Buprenorphine Treatment for Opioid Use Disorder in Community-Based Settings: Outcome Related to Intensity of Services and Urine Drug Test Results. Am J Addict. 2020 Jul;29(4):271-278. doi: 10.1111/ajad.13001. Epub 2020 Mar 11. PMID 32162434
- [Background] Wiercigroch D, Sheikh H, Hulme J. A rapid access to addiction medicine clinic facilitates treatment of substance use disorder and reduces substance use. Subst Abuse Treat Prev Policy. 2020 Jan 13;15(1):4. doi: 10.1186/s13011-019-0250-1. PMID 31931831
- [Background] Koehl JL, Zimmerman DE, Bridgeman PJ. Medications for management of opioid use disorder. Am J Health Syst Pharm. 2019 Jul 18;76(15):1097-1103. doi: 10.1093/ajhp/zxz105. PMID 31361869
- [Background] Lofwall MR, Walsh SL, Nunes EV, Bailey GL, Sigmon SC, Kampman KM, Frost M, Tiberg F, Linden M, Sheldon B, Oosman S, Peterson S, Chen M, Kim S. Weekly and Monthly Subcutaneous Buprenorphine Depot Formulations vs Daily Sublingual Buprenorphine With Naloxone for Treatment of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Intern Med. 2018 Jun 1;178(6):764-773. doi: 10.1001/jamainternmed.2018.1052. PMID 29799968
- [Background] Rosenthal RN, Ling W, Casadonte P, Vocci F, Bailey GL, Kampman K, Patkar A, Chavoustie S, Blasey C, Sigmon S, Beebe KL. Buprenorphine implants for treatment of opioid dependence: randomized comparison to placebo and sublingual buprenorphine/naloxone. Addiction. 2013 Dec;108(12):2141-9. doi: 10.1111/add.12315. Epub 2013 Sep 18. PMID 23919595
- [Background] Rosenthal RN, Lofwall MR, Kim S, Chen M, Beebe KL, Vocci FJ; PRO-814 Study Group. Effect of Buprenorphine Implants on Illicit Opioid Use Among Abstinent Adults With Opioid Dependence Treated With Sublingual Buprenorphine: A Randomized Clinical Trial. JAMA. 2016 Jul 19;316(3):282-90. doi: 10.1001/jama.2016.9382. PMID 27434441
- [Background] Ontario Drug Policy Research Network. Ontario Opioid Prescription Tool. https://odprn.ca/ontario-opioid-drug-observatory/ontario-prescription-opioid-tool/ (2018).
- [Background] Pharmacoeconomic Review Report: Buprenorphine extended-release injection (Sublocade): (Indivior Canada, Ltd.): Indication: For the management of moderate-to-severe opioid use disorder in adult patients who have been inducted and clinically stabilized on a transmucosal buprenorphine-containing product [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK546358/ PMID 31532597
- [Background] Addictions & Mental Health Ontario. Ontario Provincial Standards for Withdrawal Management Services: 2021 Standards Manual. https://amho.ca/wp-content/uploads/AMHO-Final-WMS-Ontario-Provincial-Standards-for-Withdrawal-Management-Services-September-2021-AMHO-FINAL.pdf (2021)
- [Background] Brens, C., Swoboda-Geen, C. & Gill, S. Simcoe Muskoka Opioid Strategy: An Action Plan for Our Communities. http://preventod.ca/Shared Documents/SMOS/SMOS Final Report - An Action Plan for Our Communities.pdf (2018)
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748
- [Background] McMillan DE, Gilmore-Thomas K. Stability of opioid craving over time as measured by visual analog scales. Drug Alcohol Depend. 1996 Mar;40(3):235-9. doi: 10.1016/0376-8716(96)01218-5. PMID 8861402
- [Background] Fals-Stewart W, O'Farrell TJ, Freitas TT, McFarlin SK, Rutigliano P. The timeline followback reports of psychoactive substance use by drug-abusing patients: psychometric properties. J Consult Clin Psychol. 2000 Feb;68(1):134-44. doi: 10.1037//0022-006x.68.1.134. PMID 10710848
- [Background] Reith FC, Van den Brande R, Synnot A, Gruen R, Maas AI. The reliability of the Glasgow Coma Scale: a systematic review. Intensive Care Med. 2016 Jan;42(1):3-15. doi: 10.1007/s00134-015-4124-3. Epub 2015 Nov 12. PMID 26564211
- [Background] Institute for Clinical Evaluative Sciences. Data Dictionary. ICES Data Holdings Obligations for ICES Projects https://datadictionary.ices.on.ca/Applications/DataDictionary/Default.aspx?viewmode=DataAccess (2021)
- [Background] Appropriate Use of Drug Testing in Clinical Addiction Medicine. J Addict Med. 2017 May/Jun;11 Suppl 3:1-56. doi: 10.1097/ADM.0000000000000322. No abstract available. PMID 28557842
- [Background] Dennis BB, Sanger N, Bawor M, Naji L, Plater C, Worster A, Woo J, Bhalerao A, Baptist-Mohseni N, Hillmer A, Rice D, Corace K, Hutton B, Tugwell P, Thabane L, Samaan Z. A call for consensus in defining efficacy in clinical trials for opioid addiction: combined results from a systematic review and qualitative study in patients receiving pharmacological assisted therapy for opioid use disorder. Trials. 2020 Jan 6;21(1):30. doi: 10.1186/s13063-019-3995-y. PMID 31907000
- [Background] Vernon MK, Revicki DA, Awad AG, Dirani R, Panish J, Canuso CM, Grinspan A, Mannix S, Kalali AH. Psychometric evaluation of the Medication Satisfaction Questionnaire (MSQ) to assess satisfaction with antipsychotic medication among schizophrenia patients. Schizophr Res. 2010 May;118(1-3):271-8. doi: 10.1016/j.schres.2010.01.021. Epub 2010 Feb 20. PMID 20172695
- [Background] Ling W, Nadipelli VR, Solem CT, Ronquest NA, Yeh YC, Learned SM, Mehra V, Heidbreder C. Patient-centered Outcomes in Participants of a Buprenorphine Monthly Depot (BUP-XR) Double-blind, Placebo-controlled, Multicenter, Phase 3 Study. J Addict Med. 2019 Nov/Dec;13(6):442-449. doi: 10.1097/ADM.0000000000000517. PMID 30844878
- [Background] World Health Organization. The World Health Organization Quality of Life (WHOQOL). WHOQOL BREF (2012)
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Ministry of Health & Long-Term Care. Personal Health Information Protection Act. https://www.ontario.ca/laws/statute/04p03 (2004)
- [Background] Dal-Re R, Avendano-Sola C, Bloechl-Daum B, de Boer A, Eriksson S, Fuhr U, Holm S, James SK, Mentz RJ, Perucca E, Rosendaal FR, Treweek S. Low risk pragmatic trials do not always require participants' informed consent. BMJ. 2019 Mar 27;364:l1092. doi: 10.1136/bmj.l1092. No abstract available. PMID 30917969

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05594121/Prot_SAP_000.pdf